CLINICAL TRIAL: NCT06037837
Title: Generalized Robotic Skills Assessment Using Machine Learning-Based Analysis Across Multiple Surgical Specialties
Brief Title: Improving Surgeon Performance Measures for Robot-Assisted Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-094
Record Dates: First submitted 2023-08-25; First posted 2023-09-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Surgery
Keywords: Robot assisted surgical procedure; robotic surgery; prostate surgery; kidney surgery; bladder surgery; colon surgery; pancreas surgery; gallbladder surgery; stomach surgery; uterus surgery; lung surgery; Memorial Sloan Kettering Cancer Center; 23-094
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Robotic surgeons: Participants will be robotic surgeons in urologic, gynecologic, colorectal, hepatobiliary, gastric, and thoracic surgery
  Interventions: Procedure: Robotic Surgery

INTERVENTIONS:
Procedure: Robotic Surgery — Surgeons will perform and participants will undergo robotic surgery according to the standard of care. No additional interventions will be performed on participating participants.

SUMMARY:
The purpose of this study is to develop new tools to understand surgeon performance to improve surgical training and participant outcomes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Surgeons who perform robotic surgery for candidate procedures
* Surgeons who perform candidate procedures that are frequently performed by at least three surgeons (to ensure the ability to make adequate comparisons)
* Surgeons who agree to participate in the study

Exclusion Criteria:

* Surgeons who decline to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgeons who meet the inclusion criteria will be approached by the study team for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Correlation of Automated Performance Metrics to surgeon experience | Up to 2 years
  For the primary objective, we will capture Automated Performance Metrics/APMs and will determine the association between these and other metrics and surgeon experience, which will be used to construct validation.
  APMs that will be used in the study:
  Time Metrics
  Camera Metrics
  Instrument Metrics
  System Metrics
  Articulation Metrics

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Goh, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org